CLINICAL TRIAL: NCT06335433
Title: The Dose Response Effect of Isometric Handgrip Training Frequency on Blood Pressure and Vascular Health in People With Hypertension: A Randomised Controlled Trial
Brief Title: Isometric Handgrip Training Frequency and Blood Pressure in People With Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM_30_06_22b
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Isometric Handgrip Exercise; Vascular Health; Training Frequency; Dose Response; Perceptual Responses
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Intervention Control (No Intervention): Participants will be asked to maintain their normal lifestyle patterns (i.e. diet and physical activity) and will undergo no other intervention.
- Two Sessions/Week (Experimental): Participants will complete 6-weeks of supervised isometric handgrip exercise training with a frequency of two sessions/week
  Interventions: Other: Exercise Training (Isometric Handgrip Exercise)
- Four Sessions/Week (Experimental): Participants will complete 6-weeks of supervised isometric handgrip exercise training with a frequency of four sessions/week
  Interventions: Other: Exercise Training (Isometric Handgrip Exercise)

INTERVENTIONS:
Other: Exercise Training (Isometric Handgrip Exercise) — Participants allocated to the exercise groups will complete 6 weeks of isometric handgrip exercise training (IHGT) using an electronic hand dynamometer (Camry EH101, Zhongshan Camry Electronic Co. Ltd, Guangdong) for either 2 or 4 sessions per week. Each exercise session will consist of 4 x 2-minute isometric contractions at 30% MVC with 1 minute rest periods between contractions. The first bout will be performed on the dominant arm and then the arm will be alternated for each subsequent two-minute bout. Participants will be instructed to try keep the contraction tension as close as possible to the set tension of 30% MVC using visual feedback from the dynamometer's electronic display.
  Arms: Four Sessions/Week; Two Sessions/Week

SUMMARY:
Hypertension is the most important cause of cardiovascular disease (CVD), stroke, and premature death (WHO, 2021). It is estimated by The World Health Organisation in 2021 that 1.4 billion individuals across the globe have high blood pressure, with only 14% of people actively managing these elevated levels. Simple and effective lifestyle strategies are required to help people improve their blood pressure and/or attenuate increases in blood pressure with ageing. Physical activity is one possible strategy: in previous research, several different types of physical activity have been shown to have beneficial effects on blood pressure (Blackwell et al., 2017). However, many individuals do not adhere to currently recommended levels of physical activity (150 mins of moderate intensity physical activity per week), due to a combination of the required time commitment, lack of motivation, and the associated levels of effort, exertion, and physical discomfort (Korkiakangas et al 2009). Thus, there is a need to identify alternative exercise interventions which will overcome these barriers but remain effective at improving blood pressure (Herrod, Lund, & Phillips, 2021, Toohey et al, 2018).

Low intensity isometric hand grip exercise training (IET) has been shown to result in large decreases in resting blood pressure in younger and older age groups, in both men and women, and in individuals with normal as well as elevated baseline blood pressure (Badrov et al, 2013; Bentley et al., 2018; Millar et al., 2014). In this research, IET has almost universally involved performing 4 x 2 IET holds at 30% of maximal voluntary contraction, 3 times a week, over a 4-8-week intervention (Millar et al, 2014). There are very few studies that have investigated the effect of changing different protocol parameters on changes in blood pressure and vascular health, and the minimal effective dose of IET is unknown. Defining the minimal effective dose of different types of exercise may help overcome key barriers to exercise by lowering the required time commitment, reducing perceived effort/exertion, and promoting more positive affective responses. One important modifiable parameter is training frequency and it is unknown whether reducing the frequency of IET will reduce the efficacy for improving blood pressure.

Therefore, the primary objective of this study is to determine if reducing the frequency of isometric handgrip training from four times a week to two times a week will affect the improvements in resting blood pressure and vascular health in people with hypertension. A secondary objective is to investigate the acute affective and perceptual responses to sessions of IET and the effect of training on these acute affective/perceptual responses.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years.
* Scoring low or moderate on the international physical activity questionnaire (IPAQ).
* Previous diagnosis of high blood pressure and/or a resting systolic blood pressure ≥130 but <180 mmHg (self-reported and confirmed during screening/baseline assessment).
* Currently taking no anti-hypertensive medicine or taking anti-hypertensive medicine with no treatment change within the last 4 months prior to enrollment.
* Stable dietary and physical activity patterns (including dietary supplementation) over the last 4 months

Exclusion Criteria:

* Aged <18 or >65 years
* Resting blood pressure ≥180/110 mmHg or resting heart rate >100 bpm during baseline as-sessment
* Manifest cardiovascular disease including cerebrovascular disease, heart failure, chronic kidney disease, peripheral vascular disease, or advanced retinopathy (fundus hypertonicus grades III-IV) based on a self-report health history questionnaire.
* Type 1 diabetes
* History of other chronic disease including malignancy, neurological conditions (e.g. multiple sclerosis) or respiratory conditions (e.g. COPD).
* Contraindications to exercise based on answers to the physical activity readiness questionnaire.
* Physical limitations preventing handgrip exercise (e.g. arthritis or other musculoskeletal disorder)
* Scoring "high" on the international physical activity questionnaire
* Taking more than 2 anti-hypertensive drugs or a change in treatment strategy in the previous 4 months.
* Currently taking nitrate medication (as it is commonly prescribed for angina) or on hormone replacement therapy
* Significant self-reported change in lifestyle patterns in the prior 4 months (e.g. currently on a planned diet for weight loss).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Office measured supine and seated systolic, diastolic and mean arterial pressure | 6 weeks
  Office measured supine and seated systolic, diastolic and mean arterial pressure will be measured at baseline and 3 days following the final exercise session

SECONDARY OUTCOMES:
Office measured central systolic, diastolic and mean arterial pressure | 6 weeks
  Office measured central systolic, diastolic and mean arterial pressure will be measured at baseline and 3 days following the final exercise session
24-h mean ambulatory systolic, diastolic, and mean arterial pressure | 6 weeks
  24-h mean ambulatory systolic, diastolic, and mean arterial pressure will be measured at baseline and 3 days following the final exercise session
Daytime ambulatory systolic, diastolic, and mean arterial pressure | 6 weeks
  Daytime ambulatory systolic, diastolic, and mean arterial pressure will be measured at baseline and then 3 days following the final exercise session
Sleeping ambulatory systolic, diastolic and mean arterial pressure | 6 weeks
  Sleeping ambulatory systolic, diastolic and mean arterial pressure will be measured at baseline and then 3 days after the final exercise session
Carotid-Femoral Pulse Wave Velocity | 6 weeks
  Carotid-Femoral Pulse Wave Velocity will be measured at baseline and then 3 days after the final exercise session
Affective Valence (Feeling Scale) | 6 weeks
  Affective valence will be measured at regular intervals during the isometric handgrip exercise sessions. Ratings will be collected during the first session and then during the final session of each training week.
Ratings of perceived exertion | 6 weeks
  Ratings of perceived exertion will be measured at regular intervals during the isometric handgrip exercise sessions. Ratings will be collected during the first session and then during the final session of each training week.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Metcalfe, PhD, Principal Investigator — Swansea University
Locations (1):
- Swansea University, Swansea, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No